CLINICAL TRIAL: NCT00878930
Title: Non-interventional Report on Parameters of Acceptability, Efficacy and Compliance of Fulvestrant in Post-menopausal Patients With Advanced Breast Cancer HR Positive Who Progresses to One Prior Endocrine Therapy With Antiestrogens
Brief Title: Parameters of Acceptability, Compliance and Efficacy of Fulvestrant in Post-menopausal Patients With Advance Breast Cancer
Acronym: FRAME
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sandra Mercurio / Medical Director, AZ Argentina
Other Study IDs: NIS-OAR-FAS-2008/1
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Fulvestrant; Faslodex; Acceptability; Compliance; Efficacy
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study is to obtain information of Faslodex use in the treatment of breast cancer in the clinical practice in Argentina.

DETAILED DESCRIPTION:
In Argentina, Faslodex is indicated for treating postmenopausal women with hormone receptor-positive locally advanced or metastatic breast cancer with recurrence during or after adjuvant anti-oestrogen therapy or disease progression during anti-oestrogen treatment. This study will provide information regarding the acceptability and compliance of Argentina patients to Faslodex and will provide information regarding the efficacy of this treatment in local population.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with hormone receptor-positive locally advanced or metastatic breast cancer with recurrence during or after adjuvant anti-estrogen therapy or disease progression during anti-estrogen treatment, currently receiving Faslodex
* Signature of the informed consent

Exclusion Criteria:

* Any contraindication to Faslodex administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women with advanced breast cancer hormone receptor-positive who have progressed to a one prior hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To collect real life data of acceptability and compliance on the use of Faslodex in the Argentine population. | monthly
To collect real life data of efficacy on the use of Faslodex in the Argentine population. | monthly

CONTACTS AND LOCATIONS:
Locations (16):
- Argentina (16):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Campana, Buenos Aires
  - Research Site, Ciudad de Buenos Aires, Buenos Aires
  - Research Site, La Plata, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Morón, Buenos Aires
  - Research Site, Pergamino, Buenos Aires
  - Research Site, San Martín, Buenos Aires
  - Research Site, Tandil, Buenos Aires
  - Research Site, Vicente López, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Santa Rosa, La Pampa Province
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Río Grande, Tierra del Fuego Province
  - Research Site, San Miguel de Tucumán, Tucumán Province